CLINICAL TRIAL: NCT05981300
Title: GpCRC Pediatric Gastroparesis Registry 2: Characterization and Clinical Course of Symptoms and Gastric Emptying in Pediatric, Adolescent, and Young Adult Participants With Symptoms of Gastroparesis
Brief Title: GpCRC Pediatric Gastroparesis Registry 2
Acronym: PGpR2
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Texas Tech University Health Sciences Center, El Paso (Other); Baylor College of Medicine (Other); Massachusetts General Hospital (Other); Children's Wisconsin (Unknown); Boston Children's Hospital (Other); Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 15-DK-PGpR2; U01DK112194 (NIH); U01DK112193 (NIH); U01DK074035 (NIH); U24DK074008 (NIH); IRB00416909 (Other: JHM IRB)
Record Dates: First submitted 2023-08-01; First posted 2023-08-08 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Gastroparesis; Gastroparesis-like Syndrome
Keywords: Functional Disorder of Gastrointestinal Tract; Gastro-Intestinal Disorder
MeSH Terms: conditions — Gastroparesis; Gastrointestinal Diseases; Digestive System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — Plasma and serum.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ages 8-25 with delayed gastric emptying: Participants aged 8-25 with delayed gastric emptying of solids based on gastric emptying scintigraphy
- Ages 8-25 with normal gastric emptying: Participants aged 8-25 with normal gastric emptying of solids based on gastric emptying scintigraphy

SUMMARY:
The objective of the Pediatric Gastroparesis Registry 2 is to create a national prospective registry of children, adolescents, and young adults with gastroparesis and gastroparesis-like syndrome (symptoms of gastroparesis but normal gastric emptying).

DETAILED DESCRIPTION:
An observational study to investigate the natural history and clinical course of children, adolescents, and young adults with symptoms of gastroparesis (e.g., nausea, vomiting, abdominal pain, bloating, distention) with either delayed or normal gastric emptying. To better understand these disorders, this registry will capture demographic, clinical, physiological, questionnaire, and patient outcome data to characterize the participants and their clinical course.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form and assent, as age appropriate.
* Stated willingness to comply with all study procedures and availability for the duration of the study
* 8 to 25 years of age at the time of enrollment
* Symptoms of Gp of at least 12 weeks duration: constellation of some combination of:

nausea, vomiting, early satiety, postprandial fullness; symptoms sometimes may be accompanied by upper abdominal pain

* Have undergone a gastric emptying scintigraphic study of solids using 4-hour Egg Beaters protocol (or equivalent generic liquid egg white meal) within the last 12 months who fall into one of the two categories:
* Delayed gastric emptying-defined as an abnormal 2-hour (>60% retention) and/or 4- hour (>10% retention) result based on a 4-hour scintigraphic gastric emptying study
* Gastric emptying that is not delayed but who have symptoms of Gp (designated in this study as GLS) or have previously participated in the Pediatric Gastroparesis Registry (PGpR) study
* An etiology of either diabetic or idiopathic Gp or GLS

Exclusion Criteria:

* Inability to comply with or complete the scintigraphic gastric emptying test (including allergy to eggs)
* Pregnancy
* Autism spectrum disorder, significant developmental delay, psychosis (because of inability to complete questionnaires)
* Use of narcotic analgesics greater than three days per week.
* Presence of conditions associated with GI mucosal disease (e.g., inflammatory bowel disease, known eosinophilic gastroenteritis or eosinophilic esophagitis, gastric ulcer, peptic ulcer, celiac disease)
* Presence of any other condition that could case delayed gastric emptying
* Gastrointestinal construction confirmed by upper endoscopy (EGD), upper gastrointestinal series (UGI), or abdominal CT
* Primary neurological conditions that can cause nausea and vomiting such as increased intracranial pressure, space occupying or inflammatory/infectious legions
* Acute or chronic renal failure (abnormal creatinine for age) and /or on hemodialysis or peritoneal dialysis
* Acute liver failure
* Advanced liver disease (features of portal hypertension)
* Clinically significant congenital heart disease (i.e., vaginal injury during cardiac repair)
* History of esophageal, gastric or bowel surgery.
* Metabolic disease including mitochondrial disease and inborn errors of metabolism
* Chronic lung disease (including cystic fibrosis)
* A serious chronic medical condition (e.g., inflammatory bowel disease)
* Use of medications that can affect motility during the gastric emptying study
* Any other condition, which in the option of the investigator, could explain the symptoms or could interfere with study requirements.

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will be 216 participants aged 8-25 years of age with symptoms of Gp located in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 216 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in mean symptom severity of gastrointestinal symptoms using the change in total score from the Pediatric Quality of Life Inventory (PedsQL) Gastrointestinal Symptoms Scales™ | Baseline, 48 weeks
  The PedsQL™ GI Symptoms Scales questionnaire has 65 response items covering 10 dimensions, with each item offered as a better-to-worse 5-point Likert scale choice: 0=never, 1=almost never, 2=sometimes, 3=often, 4=almost always. The item responses are transformed to a worse-to-better order and rescaled to 0-100: 0=almost always, 25= often, 50=sometimes, 75=almost never, 100= never, with higher scores indicating better health-related quality of life (HRQOL) and fewer problems or symptoms.he per-participant PedsQL™ GI Symptoms Scales total score is the sum of the 65 transformed and rescaled item responses. The primary outcome measure is the arithmetic mean of the 65 transformed item responses and is repeated at baseline and 48 weeks for each participant.

SECONDARY OUTCOMES:
Presence or absence of Carnett's sign as assessed by abdominal examination | Baseline
  Presence or absence Carnett's sign for abdominal wall pain at baseline. Carnett's sign is a finding on clinical examination in which (acute) abdominal pain remains unchanged or increases when the muscles of the abdominal wall are tensed. As part of the abdominal examination, the patient is asked to lift the head and shoulders from the examination table to tense the abdominal muscles. An alternative is to ask the patient to raise both legs with straight knees.
  A positive test indicates the increased likelihood that the abdominal wall and not the abdominal cavity is the source of the pain (for example, due to rectus sheath hematoma instead of appendicitis).
  A negative Carnett's sign is said to occur when the abdominal pain decreases when the patient is asked to lift the head; this points to an intra-abdominal cause of the pain.
Change in volume (mL) of liquid consumed as assessed by the Water Load Satiety Test | Baseline, 48 weeks
  Change from baseline to 48 weeks in amount of liquid (mL) consumed during the Water Load Satiety Test (WLST) Lower volumes are signs of impaired accommodation.
Change in Pain Catastrophizing Scale scores (PCS) | Baseline, 48 weeks
  The outcome is assessed using change in the total score at 48-weeks minus the baseline score. A negative change indicates reduced pain catastrophizing. PCS total score is computed by summing responses to all 13 items. PCS total scores range from 0 - 52.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Preidis, MD, PhD, Study Chair — Baylor College of Medicine; David Shade, JD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (6):
- United States (6):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Nationwide Children's Hospital, Columbus, Ohio
  - Texas Tech University Health Science Center, El Paso, Texas
  - Baylor College of Medicine/Texas Children's Hospital, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
The type(s) of supporting information that will be shared include deidentified individual participant data set and data dictionaries.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within 1 year of the end of the funding cycle.
Access Criteria: application
URL: https://repository.niddk.nih.gov/home

REFERENCES:
- [Background] Pasricha PJ, Grover M, Yates KP, Abell TL, Bernard CE, Koch KL, McCallum RW, Sarosiek I, Kuo B, Bulat R, Chen J, Shulman RJ, Lee L, Tonascia J, Miriel LA, Hamilton F, Farrugia G, Parkman HP; National Institute of Diabetes and Digestive and Kidney Diseases/National Institutes of Health Gastroparesis Clinical Research Consortium. Functional Dyspepsia and Gastroparesis in Tertiary Care are Interchangeable Syndromes With Common Clinical and Pathologic Features. Gastroenterology. 2021 May;160(6):2006-2017. doi: 10.1053/j.gastro.2021.01.230. Epub 2021 Feb 3. PMID 33548234
- [Background] Waseem S, Islam S, Kahn G, Moshiree B, Talley NJ. Spectrum of gastroparesis in children. J Pediatr Gastroenterol Nutr. 2012 Aug;55(2):166-72. doi: 10.1097/MPG.0b013e31824cf06e. PMID 22314391
- [Background] Rodriguez L, Irani K, Jiang H, Goldstein AM. Clinical presentation, response to therapy, and outcome of gastroparesis in children. J Pediatr Gastroenterol Nutr. 2012 Aug;55(2):185-90. doi: 10.1097/MPG.0b013e318248ed3f. PMID 22228004
- [Background] Rapkin AJ, Tsao JC, Turk N, Anderson M, Zeltzer LK. Relationships among self-rated tanner staging, hormones, and psychosocial factors in healthy female adolescents. J Pediatr Adolesc Gynecol. 2006 Jun;19(3):181-7. doi: 10.1016/j.jpag.2006.02.004. PMID 16731411
- [Background] Sizonenko PC, Aubert ML. Neuroendocrine changes characteristic of sexual maturation. J Neural Transm Suppl. 1986;21:159-81. PMID 3462329
- [Background] Angold A, Costello EJ. Depressive comorbidity in children and adolescents: empirical, theoretical, and methodological issues. Am J Psychiatry. 1993 Dec;150(12):1779-91. doi: 10.1176/ajp.150.12.1779. PMID 8238631
- [Background] Parkman HP, Yates K, Hasler WL, Nguyen L, Pasricha PJ, Snape WJ, Farrugia G, Koch KL, Abell TL, McCallum RW, Lee L, Unalp-Arida A, Tonascia J, Hamilton F; National Institute of Diabetes and Digestive and Kidney Diseases Gastroparesis Clinical Research Consortium. Clinical features of idiopathic gastroparesis vary with sex, body mass, symptom onset, delay in gastric emptying, and gastroparesis severity. Gastroenterology. 2011 Jan;140(1):101-15. doi: 10.1053/j.gastro.2010.10.015. Epub 2010 Oct 20. PMID 20965184
- [Background] Thapar N, Benninga MA, Crowell MD, Di Lorenzo C, Mack I, Nurko S, Saps M, Shulman RJ, Szajewska H, van Tilburg MAL, Enck P. Paediatric functional abdominal pain disorders. Nat Rev Dis Primers. 2020 Nov 5;6(1):89. doi: 10.1038/s41572-020-00222-5. PMID 33154368
- [Background] Camilleri M. Novel Diet, Drugs, and Gastric Interventions for Gastroparesis. Clin Gastroenterol Hepatol. 2016 Aug;14(8):1072-80. doi: 10.1016/j.cgh.2015.12.033. Epub 2016 Jan 4. PMID 26762845
- [Background] Islam S. Gastroparesis in children. Curr Opin Pediatr. 2015 Jun;27(3):377-82. doi: 10.1097/MOP.0000000000000216. PMID 25944312
- [Background] Camilleri M, Parkman HP, Shafi MA, Abell TL, Gerson L; American College of Gastroenterology. Clinical guideline: management of gastroparesis. Am J Gastroenterol. 2013 Jan;108(1):18-37; quiz 38. doi: 10.1038/ajg.2012.373. Epub 2012 Nov 13. PMID 23147521
- [Background] Pasricha PJ, Parkman HP. Gastroparesis: definitions and diagnosis. Gastroenterol Clin North Am. 2015 Mar;44(1):1-7. doi: 10.1016/j.gtc.2014.11.001. Epub 2014 Dec 24. PMID 25667018
- [Background] Lacy BE, Tack J, Gyawali CP. AGA Clinical Practice Update on Management of Medically Refractory Gastroparesis: Expert Review. Clin Gastroenterol Hepatol. 2022 Mar;20(3):491-500. doi: 10.1016/j.cgh.2021.10.038. Epub 2021 Oct 29. PMID 34757197
- [Background] Vijayvargiya P, Jameie-Oskooei S, Camilleri M, Chedid V, Erwin PJ, Murad MH. Association between delayed gastric emptying and upper gastrointestinal symptoms: a systematic review and meta-analysis. Gut. 2019 May;68(5):804-813. doi: 10.1136/gutjnl-2018-316405. Epub 2018 Jun 2. PMID 29860241
- [Background] Febo-Rodriguez L, Chumpitazi BP, Musaad S, Sher AC, Shulman RJ. Meal-Induced Symptoms in Children with Dyspepsia-Relationships to Sex and the Presence of Gastroparesis. J Pediatr. 2021 Apr;231:117-123. doi: 10.1016/j.jpeds.2020.12.048. Epub 2020 Dec 23. PMID 33359472
- [Background] Cangemi DJ, Lacy BE. Gastroparesis. Curr Opin Gastroenterol. 2021 Nov 1;37(6):596-601. doi: 10.1097/MOG.0000000000000782. PMID 34560721
- [Background] Febo-Rodriguez L, Chumpitazi BP, Shulman RJ. Childhood gastroparesis is a unique entity in need of further investigation. Neurogastroenterol Motil. 2020 Mar;32(3):e13699. doi: 10.1111/nmo.13699. Epub 2019 Aug 13. PMID 31407456
- [Background] Drossman DA, Hasler WL. Rome IV-Functional GI Disorders: Disorders of Gut-Brain Interaction. Gastroenterology. 2016 May;150(6):1257-61. doi: 10.1053/j.gastro.2016.03.035. No abstract available. PMID 27147121
- [Background] Saps M, Seshadri R, Sztainberg M, Schaffer G, Marshall BM, Di Lorenzo C. A prospective school-based study of abdominal pain and other common somatic complaints in children. J Pediatr. 2009 Mar;154(3):322-6. doi: 10.1016/j.jpeds.2008.09.047. Epub 2008 Nov 28. PMID 19038403
- [Background] Everhart JE, Ruhl CE. Burden of digestive diseases in the United States part II: lower gastrointestinal diseases. Gastroenterology. 2009 Mar;136(3):741-54. doi: 10.1053/j.gastro.2009.01.015. Epub 2009 Jan 21. No abstract available. PMID 19166855
- [Background] Everhart JE, Ruhl CE. Burden of digestive diseases in the United States part I: overall and upper gastrointestinal diseases. Gastroenterology. 2009 Feb;136(2):376-86. doi: 10.1053/j.gastro.2008.12.015. Epub 2009 Jan 3. No abstract available. PMID 19124023
- [Background] Park R, Mikami S, LeClair J, Bollom A, Lembo C, Sethi S, Lembo A, Jones M, Cheng V, Friedlander E, Nurko S. Inpatient burden of childhood functional GI disorders in the USA: an analysis of national trends in the USA from 1997 to 2009. Neurogastroenterol Motil. 2015 May;27(5):684-92. doi: 10.1111/nmo.12542. Epub 2015 Mar 22. PMID 25809794
- [Background] Mani J, Madani S, Thomas R. Economic Impact and Prognostic Factors of Functional Dyspepsia in Children. J Pediatr Gastroenterol Nutr. 2020 Apr;70(4):e65-e70. doi: 10.1097/MPG.0000000000002599. PMID 31860540
- [Background] Hyams JS, Di Lorenzo C, Saps M, Shulman RJ, Staiano A, van Tilburg M. Functional Disorders: Children and Adolescents. Gastroenterology. 2016 Feb 15:S0016-5085(16)00181-5. doi: 10.1053/j.gastro.2016.02.015. Online ahead of print. PMID 27144632
- [Background] Turco R, Russo M, Martinelli M, Castiello R, Coppola V, Miele E, Staiano A. Do Distinct Functional Dyspepsia Subtypes Exist in Children? J Pediatr Gastroenterol Nutr. 2016 Mar;62(3):387-92. doi: 10.1097/MPG.0000000000000944. PMID 26284541
- [Background] Taft TH, Doerfler B, Edlynn E, Nguyen L. The Scarcity of Literature on the Psychological, Social, and Emotional Effects of Gastroparesis in Children. Children (Basel). 2020 Aug 31;7(9):115. doi: 10.3390/children7090115. PMID 32877988
- [Background] Varni JW, Shulman RJ, Self MM, Febo-Rodriguez L, Charron H, Williams K, Nurko S, Rosen RL, Chumpitazi BP; Gastroparesis Research Consortium (GpCRC). PedsQL Gastroparesis Symptoms Module Domain and Item Development: Qualitative Methods. J Pediatr Gastroenterol Nutr. 2021 Aug 1;73(2):192-196. doi: 10.1097/MPG.0000000000003146. PMID 33853112
- [Background] Colombo JM, Deacy AD, Schurman JV, Friesen CA. Heartburn in children and adolescents in the presence of functional dyspepsia and/or irritable bowel syndrome correlates with the presence of sleep disturbances, anxiety, and depression. Medicine (Baltimore). 2021 Apr 2;100(13):e25426. doi: 10.1097/MD.0000000000025426. PMID 33787652
- [Background] Varni JW, Bendo CB, Denham J, Shulman RJ, Self MM, Neigut DA, Nurko S, Patel AS, Franciosi JP, Saps M, Yeckes A, Langseder A, Saeed S, Pohl JF. PedsQL Gastrointestinal Symptoms Scales and Gastrointestinal Worry Scales in pediatric patients with functional and organic gastrointestinal diseases in comparison to healthy controls. Qual Life Res. 2015 Feb;24(2):363-78. doi: 10.1007/s11136-014-0781-x. Epub 2014 Aug 23. PMID 25148757
- [Background] Varni JW, Bendo CB, Nurko S, Shulman RJ, Self MM, Franciosi JP, Saps M, Pohl JF; Pediatric Quality of Life Inventory (PedsQL) Gastrointestinal Symptoms Module Testing Study Consortium. Health-related quality of life in pediatric patients with functional and organic gastrointestinal diseases. J Pediatr. 2015 Jan;166(1):85-90. doi: 10.1016/j.jpeds.2014.08.022. Epub 2014 Sep 17. PMID 25241177
- [Background] Carlson MJ, Moore CE, Tsai CM, Shulman RJ, Chumpitazi BP. Child and parent perceived food-induced gastrointestinal symptoms and quality of life in children with functional gastrointestinal disorders. J Acad Nutr Diet. 2014 Mar;114(3):403-413. doi: 10.1016/j.jand.2013.10.013. Epub 2013 Dec 19. PMID 24360501
- [Background] Shava U, Srivastava A, Mathias A, Kumar N, Yachha SK, Gambhir S, Poddar U. Functional dyspepsia in children: A study of pathophysiological factors. J Gastroenterol Hepatol. 2021 Mar;36(3):680-686. doi: 10.1111/jgh.15193. Epub 2020 Aug 5. PMID 32710649
- [Background] Waseem S, Rubin L. A comprehensive review of functional dyspepsia in pediatrics. Clin J Gastroenterol. 2022 Feb;15(1):30-40. doi: 10.1007/s12328-021-01561-w. Epub 2021 Dec 2. PMID 34854065
- [Background] Pasricha PJ, Yates KP, Nguyen L, Clarke J, Abell TL, Farrugia G, Hasler WL, Koch KL, Snape WJ, McCallum RW, Sarosiek I, Tonascia J, Miriel LA, Lee L, Hamilton F, Parkman HP. Outcomes and Factors Associated With Reduced Symptoms in Patients With Gastroparesis. Gastroenterology. 2015 Dec;149(7):1762-1774.e4. doi: 10.1053/j.gastro.2015.08.008. Epub 2015 Aug 21. PMID 26299414
- [Background] Soykan I, Sivri B, Sarosiek I, Kiernan B, McCallum RW. Demography, clinical characteristics, psychological and abuse profiles, treatment, and long-term follow-up of patients with gastroparesis. Dig Dis Sci. 1998 Nov;43(11):2398-404. doi: 10.1023/a:1026665728213. PMID 9824125
- [Background] Grover M, Dasari S, Bernard CE, Chikkamenahalli LL, Yates KP, Pasricha PJ, Sarosiek I, McCallum R, Koch KL, Abell TL, Kuo B, Shulman RJ, Gibbons SJ, McKenzie TJ, Kellogg TA, Kendrick ML, Tonascia J, Hamilton FA, Parkman HP, Farrugia G. Proteomics in gastroparesis: unique and overlapping protein signatures in diabetic and idiopathic gastroparesis. Am J Physiol Gastrointest Liver Physiol. 2019 Nov 1;317(5):G716-G726. doi: 10.1152/ajpgi.00115.2019. Epub 2019 Sep 4. PMID 31482734
- [Background] Grover M, Gibbons SJ, Nair AA, Bernard CE, Zubair AS, Eisenman ST, Wilson LA, Miriel L, Pasricha PJ, Parkman HP, Sarosiek I, McCallum RW, Koch KL, Abell TL, Snape WJ, Kuo B, Shulman RJ, McKenzie TJ, Kellogg TA, Kendrick ML, Tonascia J, Hamilton FA, Farrugia G; NIDDK Gastroparesis Clinical Research Consortium (GpCRC). Transcriptomic signatures reveal immune dysregulation in human diabetic and idiopathic gastroparesis. BMC Med Genomics. 2018 Aug 7;11(1):62. doi: 10.1186/s12920-018-0379-1. PMID 30086735
- [Background] Grover M, Bernard CE, Pasricha PJ, Lurken MS, Faussone-Pellegrini MS, Smyrk TC, Parkman HP, Abell TL, Snape WJ, Hasler WL, McCallum RW, Nguyen L, Koch KL, Calles J, Lee L, Tonascia J, Unalp-Arida A, Hamilton FA, Farrugia G; NIDDK Gastroparesis Clinical Research Consortium (GpCRC). Clinical-histological associations in gastroparesis: results from the Gastroparesis Clinical Research Consortium. Neurogastroenterol Motil. 2012 Jun;24(6):531-9, e249. doi: 10.1111/j.1365-2982.2012.01894.x. Epub 2012 Feb 17. PMID 22339929
- [Background] Grover M, Farrugia G, Lurken MS, Bernard CE, Faussone-Pellegrini MS, Smyrk TC, Parkman HP, Abell TL, Snape WJ, Hasler WL, Unalp-Arida A, Nguyen L, Koch KL, Calles J, Lee L, Tonascia J, Hamilton FA, Pasricha PJ; NIDDK Gastroparesis Clinical Research Consortium. Cellular changes in diabetic and idiopathic gastroparesis. Gastroenterology. 2011 May;140(5):1575-85.e8. doi: 10.1053/j.gastro.2011.01.046. Epub 2011 Feb 4. PMID 21300066
- [Background] Friesen CA, Lin Z, Singh M, Singh V, Schurman JV, Burchell N, Cocjin JT, McCallum RW. Antral inflammatory cells, gastric emptying, and electrogastrography in pediatric functional dyspepsia. Dig Dis Sci. 2008 Oct;53(10):2634-40. doi: 10.1007/s10620-008-0207-0. Epub 2008 Mar 5. PMID 18320315
- [Background] Schurman JV, Singh M, Singh V, Neilan N, Friesen CA. Symptoms and subtypes in pediatric functional dyspepsia: relation to mucosal inflammation and psychological functioning. J Pediatr Gastroenterol Nutr. 2010 Sep;51(3):298-303. doi: 10.1097/MPG.0b013e3181d1363c. PMID 20479684
- [Background] Singh V, Singh M, Schurman JV, Friesen CA. Histopathological changes in the gastroduodenal mucosa of children with functional dyspepsia. Pathol Res Pract. 2018 Aug;214(8):1173-1178. doi: 10.1016/j.prp.2018.06.014. Epub 2018 Jun 28. PMID 30078402
- [Background] Friesen C, Singh M, Singh V, Schurman JV. An observational study of headaches in children and adolescents with functional abdominal pain: Relationship to mucosal inflammation and gastrointestinal and somatic symptoms. Medicine (Baltimore). 2018 Jul;97(30):e11395. doi: 10.1097/MD.0000000000011395. PMID 30045261
- [Background] Taki M, Oshima T, Li M, Sei H, Tozawa K, Tomita T, Fukui H, Watari J, Miwa H. Duodenal low-grade inflammation and expression of tight junction proteins in functional dyspepsia. Neurogastroenterol Motil. 2019 Oct;31(10):e13576. doi: 10.1111/nmo.13576. Epub 2019 Feb 20. PMID 30790378
- [Background] Komori K, Ihara E, Minoda Y, Ogino H, Sasaki T, Fujiwara M, Oda Y, Ogawa Y. The Altered Mucosal Barrier Function in the Duodenum Plays a Role in the Pathogenesis of Functional Dyspepsia. Dig Dis Sci. 2019 Nov;64(11):3228-3239. doi: 10.1007/s10620-019-5470-8. Epub 2019 Jan 23. PMID 30673985
- [Background] Vanheel H, Vicario M, Vanuytsel T, Van Oudenhove L, Martinez C, Keita AV, Pardon N, Santos J, Soderholm JD, Tack J, Farre R. Impaired duodenal mucosal integrity and low-grade inflammation in functional dyspepsia. Gut. 2014 Feb;63(2):262-71. doi: 10.1136/gutjnl-2012-303857. Epub 2013 Mar 8. PMID 23474421
- [Background] Neilan NA, Garg UC, Schurman JV, Friesen CA. Intestinal permeability in children/adolescents with functional dyspepsia. BMC Res Notes. 2014 May 1;7:275. doi: 10.1186/1756-0500-7-275. PMID 24886078
- [Background] McOmber ME, Ou CN, Shulman RJ. Effects of timing, sex, and age on site-specific gastrointestinal permeability testing in children and adults. J Pediatr Gastroenterol Nutr. 2010 Mar;50(3):269-75. doi: 10.1097/MPG.0b013e3181aa3aa9. PMID 20081547
- [Background] Teshima CW, Meddings JB. The measurement and clinical significance of intestinal permeability. Curr Gastroenterol Rep. 2008 Oct;10(5):443-9. doi: 10.1007/s11894-008-0083-y. PMID 18799118
- [Background] Meddings JB, Gibbons I. Discrimination of site-specific alterations in gastrointestinal permeability in the rat. Gastroenterology. 1998 Jan;114(1):83-92. doi: 10.1016/s0016-5085(98)70636-5. PMID 9428222
- [Background] Abell TL, Camilleri M, Donohoe K, Hasler WL, Lin HC, Maurer AH, McCallum RW, Nowak T, Nusynowitz ML, Parkman HP, Shreve P, Szarka LA, Snape WJ Jr, Ziessman HA; American Neurogastroenterology and Motility Society and the Society of Nuclear Medicine. Consensus recommendations for gastric emptying scintigraphy: a joint report of the American Neurogastroenterology and Motility Society and the Society of Nuclear Medicine. Am J Gastroenterol. 2008 Mar;103(3):753-63. doi: 10.1111/j.1572-0241.2007.01636.x. Epub 2007 Nov 19. PMID 18028513
- [Background] Orthey P, Dadparvar S, Parkman HP, Maurer AH. Enhanced Gastric Emptying Scintigraphy to Assess Fundic Accommodation Using Intragastric Meal Distribution and Antral Contractility. J Nucl Med Technol. 2019 Jun;47(2):138-143. doi: 10.2967/jnmt.118.215566. Epub 2018 Aug 23. PMID 30139887
- [Background] Orthey P, Yu D, Van Natta ML, Ramsey FV, Diaz JR, Bennett PA, Iagaru AH, Fragomeni RS, McCallum RW, Sarosiek I, Hasler WL, Farrugia G, Grover M, Koch KL, Nguyen L, Snape WJ, Abell TL, Pasricha PJ, Tonascia J, Hamilton F, Parkman HP, Maurer AH; NIH Gastroparesis Consortium. Intragastric Meal Distribution During Gastric Emptying Scintigraphy for Assessment of Fundic Accommodation: Correlation with Symptoms of Gastroparesis. J Nucl Med. 2018 Apr;59(4):691-697. doi: 10.2967/jnumed.117.197053. Epub 2017 Sep 28. PMID 28970332
- [Background] Piessevaux H, Tack J, Walrand S, Pauwels S, Geubel A. Intragastric distribution of a standardized meal in health and functional dyspepsia: correlation with specific symptoms. Neurogastroenterol Motil. 2003 Oct;15(5):447-55. doi: 10.1046/j.1365-2982.2003.00431.x. PMID 14507346
- [Background] Wong GK, Shulman RJ, Chiou EH, Chumpitazi BP. Decreased relative diagnostic yield of esophagogastroduodenoscopy in children with gastroparesis. J Clin Gastroenterol. 2014 Mar;48(3):231-5. doi: 10.1097/MCG.0b013e318299c8dd. PMID 23751841
- [Background] Varni JW, Bendo CB, Denham J, Shulman RJ, Self MM, Neigut DA, Nurko S, Patel AS, Franciosi JP, Saps M, Verga B, Smith A, Yeckes A, Heinz N, Langseder A, Saeed S, Zacur GM, Pohl JF. PedsQL gastrointestinal symptoms module: feasibility, reliability, and validity. J Pediatr Gastroenterol Nutr. 2014 Sep;59(3):347-55. doi: 10.1097/MPG.0000000000000414. PMID 24806837
- [Background] Velasco-Benitez CA, Gomez-Oliveros LF, Rubio-Molina LM, Tovar-Cuevas JR, Saps M. Diagnostic Accuracy of the Rome IV Criteria for the Diagnosis of Functional Gastrointestinal Disorders in Children. J Pediatr Gastroenterol Nutr. 2021 Apr 1;72(4):538-541. doi: 10.1097/MPG.0000000000003030. PMID 33394887
- [Background] Sood MR, Schwankovsky LM, Rowhani A, Zangen T, Ziring D, Furtado T, Hyman PE. Water load test in children. J Pediatr Gastroenterol Nutr. 2002 Aug;35(2):199-201. doi: 10.1097/00005176-200208000-00017. PMID 12187297
- [Background] Walker LS, Williams SE, Smith CA, Garber J, Van Slyke DA, Lipani T, Greene JW, Mertz H, Naliboff BD. Validation of a symptom provocation test for laboratory studies of abdominal pain and discomfort in children and adolescents. J Pediatr Psychol. 2006 Aug;31(7):703-13. doi: 10.1093/jpepsy/jsj062. Epub 2006 Jul 20. PMID 16861396
- [Background] Thomson H, Francis DM. Abdominal-wall tenderness: A useful sign in the acute abdomen. Lancet. 1977 Nov 19;2(8047):1053-4. doi: 10.1016/s0140-6736(77)91885-2. PMID 72957
- [Background] Carbone F, Fikree A, Aziz Q, Tack J. Joint Hypermobility Syndrome in Patients With Functional Dyspepsia. Clin Transl Gastroenterol. 2020 Nov;11(11):e00220. doi: 10.14309/ctg.0000000000000220. PMID 33259162
- [Background] Beighton P, Solomon L, Soskolne CL. Articular mobility in an African population. Ann Rheum Dis. 1973 Sep;32(5):413-8. doi: 10.1136/ard.32.5.413. No abstract available. PMID 4751776
- [Background] Smits-Engelsman B, Klerks M, Kirby A. Beighton score: a valid measure for generalized hypermobility in children. J Pediatr. 2011 Jan;158(1):119-23, 123.e1-4. doi: 10.1016/j.jpeds.2010.07.021. Epub 2010 Sep 17. PMID 20850761
- [Background] Chelimsky G, Kovacic K, Simpson P, Nugent M, Basel D, Banda J, Chelimsky T. Benign Joint Hypermobility Minimally Impacts Autonomic Abnormalities in Pediatric Subjects with Chronic Functional Pain Disorders. J Pediatr. 2016 Oct;177:49-52. doi: 10.1016/j.jpeds.2016.06.091. Epub 2016 Aug 2. PMID 27496265
- [Background] Kovacic K, Chelimsky TC, Sood MR, Simpson P, Nugent M, Chelimsky G. Joint hypermobility: a common association with complex functional gastrointestinal disorders. J Pediatr. 2014 Nov;165(5):973-8. doi: 10.1016/j.jpeds.2014.07.021. Epub 2014 Aug 20. PMID 25151198
- [Background] Juul-Kristensen B, Schmedling K, Rombaut L, Lund H, Engelbert RH. Measurement properties of clinical assessment methods for classifying generalized joint hypermobility-A systematic review. Am J Med Genet C Semin Med Genet. 2017 Mar;175(1):116-147. doi: 10.1002/ajmg.c.31540. PMID 28306223
- [Background] Remvig L, Flycht L, Christensen KB, Juul-Kristensen B. Lack of consensus on tests and criteria for generalized joint hypermobility, Ehlers-Danlos syndrome: hypermobile type and joint hypermobility syndrome. Am J Med Genet A. 2014 Mar;164A(3):591-6. doi: 10.1002/ajmg.a.36402. Epub 2014 Jan 24. PMID 24464988
- [Background] Shulman RJ, Self MM, Czyzewski DI, Goldberg J, Heitkemper M. The Prevalence of Hypermobility in Children with Irritable Bowel Syndrome and Functional Abdominal Pain Is Similar to that in Healthy Children. J Pediatr. 2020 Jul;222:134-140.e2. doi: 10.1016/j.jpeds.2020.03.033. Epub 2020 May 4. PMID 32381468
- [Background] Vera JF, Gotteland M, Chavez E, Vial MT, Kakarieka E, Brunser O. Sucrose permeability in children with gastric damage and Helicobacter pylori infection. J Pediatr Gastroenterol Nutr. 1997 May;24(5):506-11. doi: 10.1097/00005176-199705000-00002. PMID 9161942
- [Background] Sutherland LR, Verhoef M, Wallace JL, Van Rosendaal G, Crutcher R, Meddings JB. A simple, non-invasive marker of gastric damage: sucrose permeability. Lancet. 1994 Apr 23;343(8904):998-1000. doi: 10.1016/s0140-6736(94)90125-2. PMID 7909091
- [Background] Catassi C, Pierani P, Natalini G, Gabrielli O, Coppa GV, Giorgi PL. Clinical application of a simple HPLC method for the sugar intestinal permeability test. J Pediatr Gastroenterol Nutr. 1991 Feb;12(2):209-12. doi: 10.1097/00005176-199102000-00012. PMID 1904934
- [Background] Meddings JB, Sutherland LR, Byles NI, Wallace JL. Sucrose: a novel permeability marker for gastroduodenal disease. Gastroenterology. 1993 Jun;104(6):1619-26. doi: 10.1016/0016-5085(93)90637-r. PMID 8500718
- [Background] Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Med Care. 2001 Aug;39(8):800-12. doi: 10.1097/00005650-200108000-00006. PMID 11468499
- [Background] Febo-Rodriguez L, Chumpitazi BP, Musaad S, Sher AC, Varni JW, Shulman RJ. Gastrointestinal Symptoms Profile in Pediatric Patients With Gastroparesis Compared to Healthy Controls. J Pediatr Gastroenterol Nutr. 2022 Aug 1;75(2):151-158. doi: 10.1097/MPG.0000000000003484. Epub 2022 Jun 1. PMID 35653378
- [Background] Walker LS, Beck JE, Garber J, Lambert W. Children's Somatization Inventory: psychometric properties of the revised form (CSI-24). J Pediatr Psychol. 2009 May;34(4):430-40. doi: 10.1093/jpepsy/jsn093. Epub 2008 Sep 9. PMID 18782857
- [Background] Knight D, Hensley VR, Waters B. Validation of the Children's Depression Scale and the Children's Depression Inventory in a prepubertal sample. J Child Psychol Psychiatry. 1988 Nov;29(6):853-63. doi: 10.1111/j.1469-7610.1988.tb00758.x. PMID 3235493
- [Background] Claar RL, Walker LS. Functional assessment of pediatric pain patients: psychometric properties of the functional disability inventory. Pain. 2006 Mar;121(1-2):77-84. doi: 10.1016/j.pain.2005.12.002. Epub 2006 Feb 9. PMID 16480823
- [Background] Pielech M, Ryan M, Logan D, Kaczynski K, White MT, Simons LE. Pain catastrophizing in children with chronic pain and their parents: proposed clinical reference points and reexamination of the Pain Catastrophizing Scale measure. Pain. 2014 Nov;155(11):2360-7. doi: 10.1016/j.pain.2014.08.035. Epub 2014 Aug 29. PMID 25180013
- [Background] Wytiaz V, Homko C, Duffy F, Schey R, Parkman HP. Foods provoking and alleviating symptoms in gastroparesis: patient experiences. Dig Dis Sci. 2015 Apr;60(4):1052-8. doi: 10.1007/s10620-015-3651-7. Epub 2015 Apr 4. PMID 25840923
- [Background] Pilichiewicz AN, Horowitz M, Holtmann GJ, Talley NJ, Feinle-Bisset C. Relationship between symptoms and dietary patterns in patients with functional dyspepsia. Clin Gastroenterol Hepatol. 2009 Mar;7(3):317-22. doi: 10.1016/j.cgh.2008.09.007. Epub 2008 Sep 20. PMID 18929687
- [Background] Rockett HR, Breitenbach M, Frazier AL, Witschi J, Wolf AM, Field AE, Colditz GA. Validation of a youth/adolescent food frequency questionnaire. Prev Med. 1997 Nov-Dec;26(6):808-16. doi: 10.1006/pmed.1997.0200. PMID 9388792
- [Background] Chumpitazi BP, Weidler EM, Lu DY, Tsai CM, Shulman RJ. Self-Perceived Food Intolerances Are Common and Associated with Clinical Severity in Childhood Irritable Bowel Syndrome. J Acad Nutr Diet. 2016 Sep;116(9):1458-1464. doi: 10.1016/j.jand.2016.04.017. Epub 2016 Jun 15. PMID 27316779
- [Background] Revicki DA, Camilleri M, Kuo B, Szarka LA, McCormack J, Parkman HP. Evaluating symptom outcomes in gastroparesis clinical trials: validity and responsiveness of the Gastroparesis Cardinal Symptom Index-Daily Diary (GCSI-DD). Neurogastroenterol Motil. 2012 May;24(5):456-63, e215-6. doi: 10.1111/j.1365-2982.2012.01879.x. Epub 2012 Jan 27. PMID 22284754
- [Background] Parkman HP, Camilleri M, Farrugia G, McCallum RW, Bharucha AE, Mayer EA, Tack JF, Spiller R, Horowitz M, Vinik AI, Galligan JJ, Pasricha PJ, Kuo B, Szarka LA, Marciani L, Jones K, Parrish CR, Sandroni P, Abell T, Ordog T, Hasler W, Koch KL, Sanders K, Norton NJ, Hamilton F. Gastroparesis and functional dyspepsia: excerpts from the AGA/ANMS meeting. Neurogastroenterol Motil. 2010 Feb;22(2):113-33. doi: 10.1111/j.1365-2982.2009.01434.x. Epub 2009 Dec 9. PMID 20003077
- [Background] Pasricha PJ, Camilleri M, Hasler WL, Parkman HP. White Paper AGA: Gastroparesis: Clinical and Regulatory Insights for Clinical Trials. Clin Gastroenterol Hepatol. 2017 Aug;15(8):1184-1190. doi: 10.1016/j.cgh.2017.04.011. Epub 2017 Apr 12. PMID 28410896
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Grahame R, Bird HA, Child A. The revised (Brighton 1998) criteria for the diagnosis of benign joint hypermobility syndrome (BJHS). J Rheumatol. 2000 Jul;27(7):1777-9. No abstract available. PMID 10914867
- [Background] Tougas G, Eaker EY, Abell TL, Abrahamsson H, Boivin M, Chen J, Hocking MP, Quigley EM, Koch KL, Tokayer AZ, Stanghellini V, Chen Y, Huizinga JD, Ryden J, Bourgeois I, McCallum RW. Assessment of gastric emptying using a low fat meal: establishment of international control values. Am J Gastroenterol. 2000 Jun;95(6):1456-62. doi: 10.1111/j.1572-0241.2000.02076.x. PMID 10894578
- [Background] Baxter AL, Watcha MF, Baxter WV, Leong T, Wyatt MM. Development and validation of a pictorial nausea rating scale for children. Pediatrics. 2011 Jun;127(6):e1542-9. doi: 10.1542/peds.2010-1410. Epub 2011 May 29. PMID 21624874
- [Background] Varni JW, Burwinkle TM, Seid M, Skarr D. The PedsQL 4.0 as a pediatric population health measure: feasibility, reliability, and validity. Ambul Pediatr. 2003 Nov-Dec;3(6):329-41. doi: 10.1367/1539-4409(2003)0032.0.co;2. PMID 14616041
- [Background] Walker LS, Garber J, Greene JW. Psychosocial correlates of recurrent childhood pain: a comparison of pediatric patients with recurrent abdominal pain, organic illness, and psychiatric disorders. J Abnorm Psychol. 1993 May;102(2):248-58. doi: 10.1037//0021-843x.102.2.248. PMID 8315137
- [Background] Kovacs M. Rating scales to assess depression in school-aged children. Acta Paedopsychiatr. 1981 Feb;46(5-6):305-15. No abstract available. PMID 7025571
- [Background] Walker LS, Greene JW. The functional disability inventory: measuring a neglected dimension of child health status. J Pediatr Psychol. 1991 Feb;16(1):39-58. doi: 10.1093/jpepsy/16.1.39. PMID 1826329
- [Background] Parkerson HA, Noel M, Page MG, Fuss S, Katz J, Asmundson GJ. Factorial validity of the English-language version of the Pain Catastrophizing Scale--child version. J Pain. 2013 Nov;14(11):1383-9. doi: 10.1016/j.jpain.2013.06.004. Epub 2013 Sep 5. PMID 24012382
- [Background] Simren M, Mansson A, Langkilde AM, Svedlund J, Abrahamsson H, Bengtsson U, Bjornsson ES. Food-related gastrointestinal symptoms in the irritable bowel syndrome. Digestion. 2001;63(2):108-15. doi: 10.1159/000051878. PMID 11244249
- [Background] Tringali A, Balassone V, De Angelis P, Landi R. Complications in pediatric endoscopy. Best Pract Res Clin Gastroenterol. 2016 Oct;30(5):825-839. doi: 10.1016/j.bpg.2016.09.006. Epub 2016 Sep 13. PMID 27931639
- [Background] Walker LS, Caplan-Dover A, Rasquin-Weber A. Manual for the Questionnaire on Pediatric Gastrointestinal Disorders. Nashville: Vanderbilt University School of Medicine, 2000.
- [Background] Spielberger CD. Manual for the State-Trait Anxiety Inventory for Children. Palo Alto: Consulting Psychologists Press, 1973.
- [Background] PASS 2023 Power Analysis and Sample Size Software (2023). NCSS, LLC. Kaysville, Utah, USA, ncss.com/software/pass